CLINICAL TRIAL: NCT02653430
Title: Efficacy and Mechanism Study of Bariatric Surgery to Treat Moderate to Severe Obesity in Han Chinese Population
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Guang Ning, Professor, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCEMD026
Record Dates: First submitted 2015-12-30; First posted 2016-01-12 (Estimated); Last update posted 2016-04-26 (Estimated); Status verified 2016-01

CONDITIONS: Morbid Obesity
Keywords: obesity; BMI; efficacy; bariatric surgery; gut flora; fMRI
MeSH Terms: conditions — Obesity, Morbid; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bariatric Surgery (Experimental): Sleeve Gastrectomy
  Interventions: Procedure: Sleeve gastrectomy

INTERVENTIONS:
Procedure: Sleeve gastrectomy — After complete exams such as EKG，UCG，spirometry and other basic exams,estimate the condition of patient whether he(she) can tolerate a surgical operation.Then we operate the"Sleeve gastrectomy laparoscopically" by a group of experienced surgeons.

SUMMARY:
This is a long-term follow-up and interventional study in individuals who have been diagnosed with moderate to severe obesity with or without diabetes. The purpose of this study is to determine the effects of sleeve gastrectomy on weight and blood sugar control and underlying mechanisms by metabolomics, metagenomics, functional magnetic resonance imaging (fMRI) ,adipose tissue expression chip and etc.

DETAILED DESCRIPTION:
Prevalence of obesity has been increasing rapidly worldwide. Overweight and obesity prevalence surged to 35.1% according to China Noncommunicable Disease Surveillance 2010. An estimated 44% of the burden for diabetes has been attributed to these weight problems, as well as 23% and 7-41% of the burdens for ischaemic heart disease and specific cancers. So now, obesity is a very serious disease, and it is not easy to lose weight or maintain proper weight.

With the failure of non-surgical strategies, bariatric surgery has emerged as the most effective therapeutic option for the treatment of severe obesity. From the beginning, there are a lot of types of operation which have been created and then been abandoned. Now, the most common is Roux-en-Y gastric bypass, sleeve gastrectomy (SG), gastric banding, and biliopancreatic diversion. In recent years, the international status of SG surgery gradually went up. Since 2013, SG has been recommended as the preferred option of bariatric surgery by the American Weight Loss Society. However, the underlying mechanism of SG procedure is not fully clear.

In fact, clinical and translational studies over the last decade have shown that a number of gastrointestinal mechanisms, including changes in gut hormones, neural signalling, intestinal flora, bile acid and lipid metabolism can play a significant role in the effects of this procedure on energy homeostasis. This is a long-term follow-up and interventional study in individuals who have been diagnosed with moderate to severe obesity with or without diabetes. The purpose of this study is to determine the effects of SG on weight and blood sugar control and underlying mechanisms by metabolomics, metagenomics, functional magnetic resonance imaging (fMRI) ,adipose tissue expression chip and etc.

ELIGIBILITY:
Inclusion Criteria:

* BMI≥35kg/m2 with or without obesity complications
* BMI≥32kg/m2 with type 2 diabetes, high blood pressure, severe OSAHS, atherosclerotic plaque formation or other obesity complications
* Type 2 diabetes duration of ≤ 15 years, half of the lower limit of normal islet reserve function or more, C peptide ≥2.

Exclusion Criteria:

* had an operation for losing weight before
* serious hepatic or renal dysfunction
* mentally ill，serious tristimania，personality disturbance，disgnosia
* drug abuse or alcool abuse
* ulcer or tumor history or other high risks for surgery or serious gastrointestinal disease
* can not be follow-up，refuse to change the life-style
* type 1 diabetes mellitus
* self-care disable or no familial care
* obesity caused by drugs
* secondary obesity, such as monogenic obesity, obesity-related genetic syndrome, cushing syndrome and etc.

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-02; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Excess Weight Loss | up to 10 years

SECONDARY OUTCOMES:
Remission rate of type 2 diabetes mellitus or control of glycemia | up to 10 years
Waist circumference | up to 10 years
Hip circumference | up to 10 years
Fat percent determined by Inbody 720 | up to 10 years
Assessment of insulin resistance | up to 10 years
Abdominal fat deposition | up to 10 years
Apnea hypopnea index by polysomnography | up to 10 years
Appetite assessed by Three-factor eating questionnaire (TFEQ) | up to 10 years
Gut microbiome | up to 10 years
Concentration of blood metabolites | up to 10 years
Appetite signal in brain determined by fMRI | up to 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Guang Ning, MD,PhD, Principal Investigator — Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Hong J, Bo T, Xi L, Xu X, He N, Zhan Y, Li W, Liang P, Chen Y, Shi J, Li D, Yan F, Gu W, Wang W, Liu R, Wang J, Wang Z, Ning G. Reversal of Functional Brain Activity Related to Gut Microbiome and Hormones After VSG Surgery in Patients With Obesity. J Clin Endocrinol Metab. 2021 Aug 18;106(9):e3619-e3633. doi: 10.1210/clinem/dgab297. PMID 33950216
- [Derived] Chen Y, Chen L, Ye L, Jin J, Sun Y, Zhang L, Zhao S, Zhang Y, Wang W, Gu W, Hong J. Association of Metabolic Syndrome With Prevalence of Obstructive Sleep Apnea and Remission After Sleeve Gastrectomy. Front Physiol. 2021 Mar 31;12:650260. doi: 10.3389/fphys.2021.650260. eCollection 2021. PMID 33868016